CLINICAL TRIAL: NCT02022709
Title: Efficacy of Exposure and Response Prevention（ERP） and SSRIs, and Its Predictors in Obsessive-Compulsive Disorder
Brief Title: Efficacy of Exposure and Response Prevention(ERP) and SSRIs in Chinese OCD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhen Wang, Director, Research and Education Department, Shanghai Mental Health Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 124119a8601; YG2013MS65 (Other Grant/Funding Number: Biomedical Engineering Cross Project of SJTU)
Record Dates: First submitted 2013-12-15; First posted 2013-12-30 (Estimated); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Obsessive-Compulsive Disorder; Anxiety Disorders; Mental Disorders
Keywords: Cognitive Behavior Therapy; Exposure and Response/Ritual Prevention; Selective Serotonin Reuptake Inhibitors; Psychotherapy; Pharmacotherapy; Citalopram; Fluoxetine; Paroxetine; Sertraline; Fluvoxamine; fMRI; Stop Signal Task
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Mental Disorders | interventions — Fluoxetine; Sertraline; Paroxetine; Citalopram; Dexetimide; Fluvoxamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Selective Serotonin Reuptake Inhibitor (Active Comparator): In this group,routine treatment strategies will be used for patients. Any one of the SSRIs including fluoxetine, citalopram, paroxetine, sertraline, fluvoxamine ,which are approved in the treatment of OCD by SFDA, may be used for patients who are randomized to this treatment arm. The dosage depends on clinician's judgement ,but not over the maximum tolerated dosage.
  Interventions: Drug: Fluoxetine; Drug: Sertraline; Drug: Paroxetine; Drug: Citalopram; Drug: Fluvoxamine
- Exposure and Response Prevention (Active Comparator): Exposure and Response Prevention Structured protocol described by Foa et al., 2012 Patients will attend eight 1-h sessions,once a week. Benzodiazepine will be used when necessary.
  Interventions: Behavioral: Exposure and Response Prevention

INTERVENTIONS:
Drug: Fluoxetine — The dosage depends on clinician's judgement ,but not over the maximum tolerated dosage.
  Other Names: Prozac
  Arms: Selective Serotonin Reuptake Inhibitor
Drug: Sertraline — The dosage depends on clinician's judgement ,but not over the maximum tolerated dosage.
  Other Names: Zoloft
  Arms: Selective Serotonin Reuptake Inhibitor
Drug: Paroxetine — The dosage depends on clinician's judgement ,but not over the maximum tolerated dosage.
  Other Names: Seroxat
  Arms: Selective Serotonin Reuptake Inhibitor
Drug: Citalopram — The dosage depends on clinician's judgement ,but not over the maximum tolerated dosage.
  Other Names: Cipramil
  Arms: Selective Serotonin Reuptake Inhibitor
Drug: Fluvoxamine — The dosage depends on clinician's judgement ,but not over the maximum tolerated dosage.
  Other Names: Luvox
  Arms: Selective Serotonin Reuptake Inhibitor
Behavioral: Exposure and Response Prevention — 8 exposure and response prevention (ERP) sessions,once a week
  Other Names: Exposure and Rituals Prevention
  Arms: Exposure and Response Prevention

SUMMARY:
The purpose of this study is to evaluate the efficiency of SSRIs（Selective Serotonin Reuptake Inhibitor） ,ERP（Exposure and Response Prevention） and the combination of the two therapies for OCD(Obsessive-Compulsive Disorder) patients ,at the same time, to find out the biological or psychological predictors of treatment response in Chinese population.

DETAILED DESCRIPTION:
Although Selective Serotonin Reuptake Inhibitors(SSRIs) and Cognitive Behavior Therapy (CBT) including Exposure and Response Prevention(ERP) are two kinds of the first line treatments for OCD(Obsessive-Compulsive Disorder) according to APA（American Psychological Association）guideline. Both of the treatments are effective, but few research has been done to find out who are more responsive to one treatment than the other. The aim of our research is to evaluate the efficiency of SSRIs ,ERP and the combination of the two therapies for OCD patients ,at the same time, to find out the biological and psychological predictors of treatment response in Chinese population.

This is a randomized, single-blind, cross-over design study.Approximately 60 patients will be randomized to SSRIs or ERP group. Neuropsychological assessment and fMRI(Functional Magnetic Resonance Imaging） will be performed at baseline,during the treatment and at the end of the study. The research has two period. In the first period(before week 8) ,the patients will have monotherapy. In the second period(after week 8), rates of improvement based on the YBOCS(Yale-Brown Obsessive Compulsive Scale) scores will be assessed. The patient will be considered responsive to treatment when he or she has a reduction in YBOCS score ≥ 35% of the score at the baseline.If the patient is responsive to the treatment that he or she has received at the first 8 weeks,he or she will continue to follow the previous treatment strategy.If not,the patient will have a combination of SSRIs and ERP treatment for another 8 weeks. The follow-up period will last up to 6 months.The result of the study will improve our knowledge about the efficacy of the two first line treatments .Also,it will help us to find out the predictors of the outcome of the two different kinds of treatments.Strategy of clinical treatment of OCD will be more individualized in the future.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with primary OCD as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-) criteria;Cleaning or checking as primary OCD symptoms
* Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) score of ≥ 16
* Never receiving adequate treatment or stop receiving treatment for at least 8 weeks
* Having an education degree of high school or above
* Accepting to participate in the study

Exclusion Criteria:

* Having significant medical illnesses that would interfere with the conduct of the study
* Clinically significant abnormal laboratory finding
* Having comorbid psychiatric conditions according to the criteria set forth in the DSM-IV(administered by the Mini-International Neuropsychiatric Interview (MINI))
* The current OCD symptoms are too severe that the patient cannot finish the evaluation or receive the ERP
* Being currently at risk for suicide
* Being pregnant or having the intention to be pregnant before the end of the study
* A history of having inadequate response to adequate SSRIs or CBT treatment
* Subjects who are unable to undergo the MRI

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-01; Primary Completion 2017-11-18 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
The change of Yale-Brown Obsessive-Compulsive Scale score | from baseline to month 6
  Patients were assessed at 0 week(w), 2w, 4w, 8w, 10w, 12w, 16w(0 month), 6 month

SECONDARY OUTCOMES:
The change of Beck Depression Inventory(BDI) score | from baseline to month 6
  Patients were assessed at 0 week(w), 2w, 4w, 8w, 10w, 12w, 16w(0 month), 6 month
The change of Beck Anxiety Inventory(BAI) score | from baseline to month 6
  Patients were assessed at 0 week(w), 2w, 4w, 8w, 10w, 12w, 16w(0 month), 6 month
The change of Stress Perceived Questionnaire (PSS-10) score | from baseline to month 6
  Patients were assessed at 0 week(w),16w(0 month), 6 month
The change of Behavioral Inhibition/Behavioral Activation System Scales score | from baseline to month 6
  Patients were assessed at 0 week(w), 16w(0 month), 6 month
The change of Barratt Impulsiveness Scale 11 (BIS-11) score | from baseline to month 6
  Patients were assessed at 0 week(w), 16w(0 month), 6 month
The change of Obsessive Beliefs Questionnaire-44(OBQ-44) score | from baseline to month 6
  Patients were assessed at 0 week(w), 16w(0 month), 6 month
The NEO-Five Factor Inventory-Revised (NEO-FFI-R) | at baseline
  Patients were assessed at 0 week(w),
The Early Trauma Inventory Self Report-Short Form(ETISR-SF) | at baseline
  Patients were assessed at 0 week(w)

OTHER OUTCOMES:
Stop Signal Task (SST) | from baseline to month 6
  a measure of behavioral response inhibition
fMRI(Functional Magnetic Resonance Imaging) - stop signal task | from baseline to month 6
  a measure of behavioral response inhibition
C Reaction Protein(CRP) | from baseline to month 6
  for safety considerations
Complete Blood Count | from baseline to month 6
  for safety considerations
Liver and Kidney Function | from baseline to month 6
  for safety considerations
Resting State Functional Magnetic Resonance Imaging | from baseline to month 6
  to quantify brain network

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, Ph.D, M.D, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China